CLINICAL TRIAL: NCT01810302
Title: Intraventricular Nicardipine for the Treatment of Cerebral Vasospasm: Prospective Pilot Study
Brief Title: Safety Study of Nicardipine to Treat Cerebral Vasospasm
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to secure drug.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 034-2013
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Cerebral Vasospasm
Keywords: Vasospasm; Subarachnoid hemorrhage; Aneurysmal subarachnoid hemorrhage; Nicardipine; Intrathecal; SAH; aSAH
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage | interventions — Nicardipine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicardipine hydrochloride (Experimental): Nicardipine hydrochloride 4mg by intrathecal administration twice a day until post-hemorrhage day 10.
  Interventions: Drug: Nicardipine hydrochloride
- Preservative-free normal saline (Placebo Comparator): Preservative-free normal saline 1.6 mL by intrathecal administration twice a day until post-hemorrhage day 10.
  Interventions: Drug: Preservative-free normal saline

INTERVENTIONS:
Drug: Nicardipine hydrochloride — Nicardipine hydrochloride 4mg by intrathecal administration twice a day until post-hemorrhage day 10.
  Other Names: Nicardipine; Cardene
  Arms: Nicardipine hydrochloride
Drug: Preservative-free normal saline — Preservative-free normal saline 1.6 mL by intrathecal administration twice a day until post-hemorrhage day 10.
  Other Names: Normal saline; Placebo; NS
  Arms: Preservative-free normal saline

SUMMARY:
The purpose of this study is to determine if intrathecal nicardipine is safe for the treatment of cerebral vasospasm.

DETAILED DESCRIPTION:
Subarachnoid hemorrhage accounts for approximately 5% of all strokes and affects 30,000 Americans per year. Poor outcome from aneurysmal subarachnoid hemorrhage (SAH) occurs in 50 to 75% of patients, and this is attributed to secondary ischemia in approximately 30% of patients. This delayed cerebral ischemia has been attributed to the anatomic narrowing of arteries in the cerebral vasculature which occurs following SAH.

Because of this relationship between cerebral vasospasm, cerebral ischemia, and poor outcome, there has been significant effort to establish treatments that decrease the incidence of vasospasm after SAH. Currently, medications and hemodynamic maneuvers are used as standard of care for the treatment of vasospasm and to improve outcome after SAH.

The calcium channel blocker, nimodipine, is one of the few treatments for vasospasm that has been shown to be of proven benefit. Nicardipine is another calcium channel blocker that has been evaluated in several studies via an intravenous administration route. These studies did show significant improvements in symptomatic and angiographic vasospasm, although a benefit in outcome was not seen. However, the intravenous administration of nicardipine was associated with significant systemic side effects that may have affected outcome including hypotension, pulmonary edema, and azotemia.

The administration of nicardipine via an intrathecal route avoids the systemic complications associated with intravenous dosing since the direct cerebrospinal fluid dosing is much lower. The result is that the systemic concentration will remain low avoiding systemic side effects, and central nervous system concentration will remain high. We propose that this difference may improve outcomes while minimizing complication related effects on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age and older
* Subarachnoid hemorrhage documented on head CT
* Fisher Grade 3 or 4
* Hunt Hess Grade 1-5
* Cerebral aneurysm as definitive source of subarachnoid hemorrhage
* Cerebral aneurysm must be treated via open or endovascular techniques
* Presence of external ventricular drain
* Written informed consent obtained from subject or subject's legally authorized representative

Exclusion Criteria:

* Absence or inability to have an external ventricular drain (coagulopathy)
* Non-aneurysmal subarachnoid hemorrhage (perimesencephalic)
* Untreated cerebral aneurysm
* Inability to be randomized prior to post-hemorrhage day 4
* Elevated intra-cranial pressures that would preclude external ventricular drain clamping for 30-60 minutes
* Inability to administer study medication (severe intra-ventricular hemorrhage, occluded external ventricular drain)
* Inability to obtain angiography (coagulopathy, renal failure)
* Pregnant
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spiros L. Blackburn, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicardipine Hydrochloride | Preservative-free Normal Saline
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Death | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicardipine Hydrochloride | Preservative-free Normal Saline | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bacterial Meningitis.
Time Frame: Day 1 of study drug until post-hemorrhage day 10.
Population: Number of participants were not sufficient to perform data analysis.
Arm/Group | Nicardipine Hydrochloride | Preservative-free Normal Saline
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Cerebral Vasospasm.
Time Frame: Day 1 of study drug until post-hemorrhage day 10.
Population: Number of participants were not sufficient to perform data analysis.
Arm/Group | Nicardipine Hydrochloride | Preservative-free Normal Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event monitoring began at the initiation of study procedures and continued until post-hemorrhage day 17.
Arm/Group | Nicardipine Hydrochloride | Preservative-free Normal Saline
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nicardipine Hydrochloride (N=1) | Preservative-free Normal Saline (N=1)
Intracranial Hemorrhage (Nervous system disorders) | 1 | 0
Gastointestinal Bleed (Gastrointestinal disorders) | 1 | 0
Gastic Ulcer Perforation (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nicardipine Hydrochloride (N=1) | Preservative-free Normal Saline (N=1)
Altered Mental Status (Nervous system disorders) | 1 | 1
Fever (General disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Cerebrospinal Fluid Leakage (Nervous system disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Thromboembolic Event (Vascular disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This single center study was terminated early due to inability to maintain an adequate drug supply; therefore, statistical analysis of the 2 participants was not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes